CLINICAL TRIAL: NCT01448421
Title: A Prospective, Single Arm Feasibility Study to Evaluate the Safety and Performance of the Keystone Heart Embolic Deflection Device in Patients Undergoing Transcatheter Aortic Valve Replacement (TAVR)
Brief Title: DEFLECT I: Keystone Heart Embolic Deflection Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keystone Heart (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DEFLECT I
Record Dates: First submitted 2011-09-20; First posted 2011-10-07 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2014-01

CONDITIONS: Aortic Stenosis
Keywords: TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Keystone Heart Embolic Deflection Device (Experimental): Protected Transcatheter Aortic Valve Replacement
  Interventions: Device: Keystone Heart Embolic Deflection Device

INTERVENTIONS:
Device: Keystone Heart Embolic Deflection Device — The Keystone Heart Embolic Deflection Device is used in the aortic arch to deflect and to reduce embolic material (debris/thrombus) to the cerebral/carotid arteries during endovascular procedures.

SUMMARY:
This is a research study using the Keystone Heart Embolic Deflection Device and involving patients with aortic stenosis (a disease of the aortic valve), to be treated with Transcatheter Aortic Valve Replacement (TAVR).

The TAVR procedure consists in replacing the diseased aortic valve by a new artificial valve. The new valve is put into place using a long, thin tube called a catheter that is inserted into a small incision (cut) in the patient's groin and threaded through his/her arteries up to the heart.

DETAILED DESCRIPTION:
This is a research study using the Keystone Heart Embolic Deflection Device and involving patients with aortic stenosis (a disease of the aortic valve), to be treated with Transcatheter Aortic Valve Replacement (TAVR).

The TAVR procedure consists in replacing the diseased aortic valve by a new artificial valve. The new valve is put into place using a long, thin tube called a catheter that is inserted into a small incision (cut) in the patient's groin and threaded through his/her arteries up to the heart.

During the TAVR procedure, there is a risk that an abnormal particle (called embolism) could break off from inside the arteries and travel to the brain. The embolism could be made of clumps of blood (clots), air, part of your body tissue, or part of a medical device. If the embolism is carried through the blood to the brain, it could cause a stroke or other neurological (brain) problems. A stroke happens when blood flow to a part of the brain is blocked, causing brain cells to die.

The Keystone Heart Embolic Deflection Device has been developed to prevent an embolism from going to the brain and causing a stroke or other brain damage. The device is a wire mesh filter that covers the vessels that carry blood to brain, deflecting any any blood clots or other materials away from the patient's brain and towards the lower body, where they are less likely to cause harm.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 years of age.
2. Patient meets indications for TAVR procedure.
3. The patient is willing to comply with protocol-specified follow-up evaluations.
4. The patient, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Medical Ethics Committee or Institutional Review Board.

Exclusion Criteria:

1. Patients undergoing TAVR via the trans-axillary, subclavian, or direct aortic route
2. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to index procedure per site standard test.
3. Patients with known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure (according to definition) or AMI >72 hours preceding the index procedure, in whom creatine kinase and creatine kinase have not returned to within normal limits at the time of procedure.
4. Patients who are currently experiencing clinical symptoms consistent with new onset AMI, such as nitrate-unresponsive prolonged chest pain.
5. Patients with impaired renal function (estimated Glomerular Filtration Rate [estimated Glomerular Filtration Rate] <30, calculated from serum creatinine by the Cockcroft-Gault formula)
6. Patients with a platelet count of <100.000 cells/mm³ or > 700.000 cells/mm³ or a white blood cell < 3000 cells/mm³ within 7 days prior to index procedure.
7. Patients with a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated, or who will refuse transfusion.
8. Patients who have received any organ transplant or are on a waiting list for any organ transplant.
9. Patients with known other medical illness or known history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation or is associated with a life expectancy of less than one year.
10. Patients with known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, nitinol, stainless steel alloy, and/or contrast sensitivity that cannot be adequately pre-medicated.
11. Patients with a history of a stroke or transient ischemic attack (TIA) within the prior 6 months.
12. Patients with an active peptic ulcer or history of upper gastrointestinal (GI) bleeding within the prior 6 months.
13. Patients presenting with cardiogenic shock.
14. Patients with severe peripheral arterial disease that precludes 9 French sheath vascular access.
15. Patients with documented friable or mobile atherosclerotic plaque in the aortic arch.
16. Patients with contraindication to cerebral MRI.
17. Patients who have a planned treatment with any other investigational device or procedure during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mullen, Md., Principal Investigator — The Heart Hospital, London, UK

REFERENCES:
- [Derived] Baumbach A, Mullen M, Brickman AM, Aggarwal SK, Pietras CG, Forrest JK, Hildick-Smith D, Meller SM, Gambone L, den Heijer P, Margolis P, Voros S, Lansky AJ. Safety and performance of a novel embolic deflection device in patients undergoing transcatheter aortic valve replacement: results from the DEFLECT I study. EuroIntervention. 2015 May;11(1):75-84. doi: 10.4244/EIJY15M04_01. PMID 25868876

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Keystone Heart Embolic Deflection Device
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: all baseline characteristics were provided for study participants
Arm/Group | Keystone Heart Embolic Deflection Device
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 13
Region of Enrollment [Number; unit: participants]
  Netherlands | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Where the Device Accessed, Deployed and Was Positioned in the Aortic Arch (Device Performance)
Description: Device ability to access and deploy in the aortic arch and position the device to cover all three vessels.
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Keystone Heart Embolic Deflection Device
Number analyzed (Participants) | 37
Participants | 33

2. Primary Outcome: Number of Serious Adverse Events Related to Investigational Device and Procedure
Description: Incidence of investigational device- and investigational procedure-related serious adverse events
Time Frame: 30 days follow-up
Measure: Number; unit: serious adverse events
Arm/Group | Keystone Heart Embolic Deflection Device
Number analyzed (Participants) | 37
serious adverse events | 0

ADVERSE EVENTS:
Arm/Group | Keystone Heart Embolic Deflection Device
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon completion of the Clinical Trial the Principal Investigator and Sponsor shall co-operate in producing a report of the Clinical Trial. The Sponsor will provide the Institution and/or Principal Investigator with the necessary results, and the Institution and/or Principal Investigator will be authorized to publish the results.